CLINICAL TRIAL: NCT07381153
Title: Cytotoxicity Evaluation of INOX (Nanoksa G Plus) High-Performance Polymer Discs on Cell Cultures: An In-Vitro Experimental Study
Brief Title: In-Vitro Cytotoxicity Assessment of INOX (Nanoksa G Plus) Polymer Discs
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer of Periodontology, Faculty of Dentistry, Cairo University , Cairo, Egypt, Cairo University
Other Study IDs: 12l2025
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cytotoxicity
Keywords: INOX; Nanoksa G Plus; INVITRO

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the cytotoxicity of INOX (Nanoksa G Plus) high-performance polymer discs on cell cultures using standardized in-vitro assays. The primary objective is to assess cell viability after exposure to INOX extracts. Secondary objectives include examining cell membrane integrity, cellular morphology, comparing effects across extract concentrations, and determining whether INOX meets accepted non-cytotoxicity standards.

ELIGIBILITY:
Inclusion Criteria:

To assess cell viability following exposure to INOX material extracts using a quantitative cell viability assay.

Exclusion Criteria:

To evaluate cell membrane integrity following exposure to INOX extracts. To assess cellular morphology after exposure to the material. To compare cytotoxic effects at different extract concentrations. To determine whether INOX meets accepted non-cytotoxicity thresholds.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Invitro study to evaluate the cytotoxicity of INOX (Nanoksa G Plus) high-performance polymer discs on cell cultures using standardized in-vitro assays.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Cell viability | JANUARY 2026
  Cell viability, assessed using a quantitative assay (MTT, XTT, or Alamar Blue).